CLINICAL TRIAL: NCT01198015
Title: Metabolic Evaluation of Nutrition in Rett Syndrome: Creatine Metabolism
Brief Title: Creatine Metabolism in Rett Syndrome
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Prof. dr. L.M.G. Curfs, Maastricht University Medical Center
Other Study IDs: NL32481.068.10; MEC-10-2-038 (Other: Medical Ethical Committee University Hospital Maastricht)
Record Dates: First submitted 2010-09-02; First posted 2010-09-09 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2011-02

CONDITIONS: Rett Syndrome
Keywords: Rett syndrome; Nutritional status; Creatine metabolism
MeSH Terms: conditions — Rett Syndrome

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, serum, leucocytes, erythrocytes, fibroblasts.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rett syndrome girls: The study population (identical to the population in the preliminary research project) consists of a well-defined group of thirteen Dutch RTT girls with complete clinical, molecular, neurophysiological and metabolic work-up.

SUMMARY:
Rett syndrome (RTT) is an X-linked severe neurodevelopmental disorder. Despite their good appetite, many females with RTT meet the criteria for moderate to severe malnutrition. The pathological mechanism is barely understood. Although feeding difficulties may play a role in this, other constitutional factors as altered metabolic processes are suspected. Preliminary research showed elevated plasma creatine concentrations and increased urinary creatine/creatinine ratios in half of the RTT girls.

The aim of this study is to confirm previous findings and examine the functionality of the creatine transporter in RTT girls.

The investigators assume that previous findings will be confirmed, and are due to an altered functionality of the creatine transporter.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of RTT (meeting consensus diagnostic criteria (Hagberg et al, 2002));
* MECP2-mutation;
* Complete neurophysiological work-up;
* Participant preliminary research (research protocol NL25356.068.08).

Exclusion Criteria:

* Male gender

Ages: 3 Years to 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population (identical to the population in the preliminary research project) consists of a well-defined group of thirteen Dutch RTT girls with complete clinical, molecular, neurophysiological and metabolic work-up.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Confirm previous findings and examine the functionality of the creatine transporter in RTT girls | One hour
  Blood as well as urine samples will be collected to confirm previous findings concerning plasma and urine creatine concentrations. Furthermore, blood samples will be used to perform mutation analysis of the SCL6A8 gene. Secondary, a skin biopsy will be collected for functional studies regarding the creatine transporter in RTT girls. By comparing intracellular and extracellular creatine concentrations, one can assess the functionality of the creatine transporter.

CONTACTS AND LOCATIONS:
Overall Officials: Leopold MG Curfs, Professor, Study Director — Maastricht University Medical Center; Eric EJ Smeets, MD, Study Director — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands